CLINICAL TRIAL: NCT01987830
Title: A Study to Evaluate Vascular Normalization in Patients With Recurrent Glioblastoma Treated With Bevacizumab Using [11C]Temozolomide PET and Vascular MRI
Brief Title: Bevacizumab w / Temozolomide PET & Vascular MRI For GBM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Gerstner, MD, Principal Investigators, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 13-322
Record Dates: First submitted 2013-11-13; First posted 2013-11-19 (Estimated); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Recurrent Glioblastoma
Keywords: Recurrent glioblastoma
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TMZ-PET scans/ MRI-PET Scan (Other): The investigators plan to study patients with recurrent glioblastoma whose clinical care plan includes treatment with bevacizumab and temozolomide. Patients taking daily temozolomide 50 mg/m2/day will undergo a PET scan using radiolabeled temozolomide (TMZ-PET) at 3 time points: 7-13 days after initiation of temozolomide but before beginning bevacizumab ("baseline"- temozolomide steady-state scan), 1 day after initiation of bevacizumab (day 15) and 1 month after initiation of bevacizumab (day 45). Arterialized venous blood samples will be collected during the imaging in order to measure radioactivity, blood metabolites, and the relationship between radiotracer uptake and tumor features such as blood-brain barrier (BBB) breakdown and tumor blood flow.
  In addition, we will explore the link between flow, permeability, and tumor temozolomide retention. These studies will be performed using our human simultaneous MRI-PET imaging camera.
  Interventions: Device: MRI-PET; Device: TMZ-PET

INTERVENTIONS:
Device: MRI-PET — * [11C] temozolomide for PET scan and a contrast dye for the MRI scan
  * Drawing blood to assess the radioactivity of [11C] temozolomide
Device: TMZ-PET — The PET scan will take approximately 90 minutes. You will receive one injection of [11C] temozolomide. Following the injection of the radioactive substance, blood samples will be taken from the second IV line.

SUMMARY:
This research study is exploring how the blood vessels in the participant's tumor change from treatment with bevacizumab, and how these changes affect the way their tumor absorbs temozolomide (TMZ).

The pilot part of this study is to evaluate the use of [11C] temozolomide PET (TMZ-PET) scans and MRI scans to tell investigators more about how standard treatment with bevacizumab affects the blood vessels in the participant's tumor, and how these changes affect the way the participant's tumor absorbs temozolomide. "Investigational" means that the role of TMZ-PET scans is still being studied and that research doctors are trying to find out more about it.

Bevacizumab is approved by the U.S. Food and Drug Administration for use in people with the participant's type of cancer. It works by blocking signals on a specific protein called vascular endothelial growth hormone (VEGF), which plays a role in promoting the growth of spread of tumor blood vessels. Bevacizumab is an "anti-VEGF' agent because it is designed to slow the growth of the participant's cancer.

Since anti-VEGF agents also affect normal blood vessels in the brain, they can inhibit the way other drugs used in combination with bevacizumab are delivered to the tumor. Researchers are looking for how bevacizumab affects delivery of chemotherapy, in this case temozolomide.

In PET scans, a radioactive substance is injected into the body. The scanning machine finds the radioactive substance, which tends to go to cancer cells.

For the PET scans in this research study, the investigators are using a radioactive substance called [11C] temozolomide, which is chemically identical to the prescription drug TMZ. TMZ is FDA approved as a chemotherapeutic agent in cancer but [11C] temozolomide is an investigational agent.

In this research study, participants will receive standard treatment with bevacizumab and oral temozolomide as well as standard MRI scans. In addition, participants will undergo TMZ-PET scans before and after treatment with bevacizumab. The first TMZ-PET scan will occur 7-13 days after starting treatment with oral temozolomide but before beginning treatment with bevacizumab, day 1 after starting treatment with bevacizumab and 1 month after starting bevacizumab. TMZ-PET scans will be given at the same time as a vascular MRI, which will evaluate the changes in tumor blood flow, blood volume, and how receptive blood vessels are while also measuring how much TMZ is in the brain.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing the consent form, the participant will be asked to undergo some screening tests or procedures to find out if they can be in the research study. Many of these tests and procedures are likely to be part of regular cancer care and may be done even if it turns out that the participant does not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about the participant's health, current medications, and any allergies.
* Physical Exam including measuring the participant's height, weight, and vital signs
* Performance status, which evaluates how the participant is able to carry on with your usual activities.
* Blood tests.
* Blood pregnancy test for women of childbearing potential
* Urine test.

If these tests show that the participant is eligible to participate in the research study, the participant will begin the study treatment. If the participant does not meet the eligibility criteria, the participant will not be able to participate in this research study.

After the screening procedures confirm that the participant is eligible to participate in the research study:

Please note that this study does not add any additional treatment to participants with your type of cancer. There will be no change in your treatment with bevacizumab and daily temozolomide based on the results of any procedures or tests carried out as a part of the study.

Before each set of scans the participant will have the following tests and procedures:

* Routine blood tests to check the participant's overall health
* Creatinine clearance blood test to check for proper kidney function
* Blood pregnancy test for women of childbearing potential

After the participant have been taking oral TMZ for 7-13 days, the participant will have:

- An assessment of their tumor by DCE-MRI (Dynamic Contrast Enhanced-Magnetic Resonance Imaging) scans and PET (Positron Emission Tomography) scan

MRI-PET Scan Procedure:

The participant will have their scans performed in Charlestown, MA at the Martinos Center. The participant will be injected with two separate intravenous (IV) lines for:

* [11C] temozolomide for PET scan and a contrast dye for the MRI scan
* Drawing blood to assess the radioactivity of [11C] temozolomide [11C] temozolomide PET Scans (TMZ PET Scan):
* The PET scan will take approximately 90 minutes. The participant will receive one injection of [11C] temozolomide. Following the injection of the radioactive substance, blood samples will be taken from the second IV line.

MRI Scan:

- MRI scans will last about 60-75 minutes. This will occur at the same time as the PET scan. The participant will be injected with contrast dye twice during the MRI scan.

The MR-PET scan(s) will be performed again on Day 1 after initiation of bevacizumab (or Day 15 after initiation of temozolomide) and Day 30 after initiation of bevacizumab (on Day 45 after initiation of temozolomide).

Blood samples will be collected during both scans in order to measure how your blood vessels are processing the radiotracer [11C] temozolomide and how well it is being delivered to the tumor tissue. Blood samples will be drawn 2.5, 5, 10, 20, 40, 60, 75, and 90 minutes after the [11C] temozolomide injection.

The participant will be assessed for side effects via clinic visit or phone call about 24 hours after each of the visits above.

- Planned Follow-up: The investigators would like to call the participant every 3 months for three years after their second MR-PET scan to see how they are doing and if the participant is experiencing any side effects. If the participant was removed from the study due to an unacceptable side effect, the participant will be followed until it has been resolved.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must have histologically confirmed glioblastoma and evidence of recurrence > 2 months since last cycle of temozolomide. Patients with low-grade tumors who have progressed to glioblastoma are eligible.
* Patients must have received at least 6 months of monthly temozolomide previously.
* Participants must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as > 10 mm. See section 10 for the evaluation of measureable disease.
* Only patients for whom their neuro-oncologist has planned to give bevacizumab and temozolomide 50mg/m2/day as part of their treatment are eligible for this study
* Age > 18 years. Because no dosing or adverse event data are currently available on the use of radiolabeled temozolomide in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric trials.
* Life expectancy of greater than 3 months.
* Karnofsky performance status > 60 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,000/mcL
* Platelets > 100,000/mcL
* total bilirubin within normal institutional limits
* AST (SGOT)/ALT (SGPT) < 2.5 X institutional upper limit of normal
* creatinine within normal institutional limits or creatinine clearance > 60 mL/min/1.73 m2 for subjects with creatinine levels about institutional normal .
* Patient must be able to undergo MRI and PET scans.
* Patients must be maintained on a stable corticosteroid regimen for 5 days prior each MR-PET scan.
* The effects of radiolabeled temozolomide on the developing human fetus are unknown. For this reason and because radiopharmaceuticals agents are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to temozolomide.
* Participants who have already received anti-VEGF or experimental anti-angiogenic therapy for glioblastoma.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because radiolabeled temozolomide is a radiopharmaceutical agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with radiopharmaceutical agents, breastfeeding should be discontinued if the mother is treated with radiopharmaceutical agents. These potential risks may also apply to other agents used in this study.
* HIV-positive individuals on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with radiolabeled temozolomide. In addition, these individuals are at increased risk of lethal infections when treated with marrow-suppressive therapy. Appropriate studies will be undertaken in participants receiving combination antiretroviral therapy when indicated.
* Patients who are no suitable to undergo MRI or use gadolinium contrast due to:
* Claustrophobia
* Presence of metallic objects or implanted medical devices in body (i.e. cardiac pacemaker, aneurysm clips, surgical clips, prostheses, artificial hearts, valves with steel parts, metal fragments, shrapnel, tattoos near the eye, or steel implants)
* Sickle cell disease
* Renal failure
* Reduced renal function, as determined by creatinine clearance < 30 mL/min based on a serum creatinine level obtained within 28 days prior to registration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11; Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Gerstner, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachuesett General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TMZ-PET Scans/ MRI-PET Scan: Patients taking daily temozolomide 50 mg/m2/day will undergo a PET scan using radiolabeled temozolomide (TMZ-PET) at 3 time points: 7-13 days after initiation of temozolomide but before beginning bevacizumab ("baseline"- temozolomide steady-state scan), 1 day after initiation of bevacizumab (day 15) and 1 month after initiation of bevacizumab (day 45). Arterialized venous blood samples were collected during the imaging in order to measure radioactivity, blood metabolites, and the relationship between radiotracer uptake and tumor features such as blood-brain barrier (BBB) breakdown and tumor blood flow.
Period: Overall Study
Arm/Group | TMZ-PET Scans/ MRI-PET Scan
Started | 13
Completed | 12
Not Completed | 1
Not completed — Never received baseline scan | 1

BASELINE CHARACTERISTICS:
Groups:
- TMZ-PET Scans/ MRI-PET Scan: The investigators plan to study patients with recurrent glioblastoma whose clinical care plan includes treatment with bevacizumab and temozolomide. Patients taking daily temozolomide 50 mg/m2/day will undergo a PET scan using radiolabeled temozolomide (TMZ-PET) at 3 time points: 7-13 days after initiation of temozolomide but before beginning bevacizumab ("baseline"- temozolomide steady-state scan), 1 day after initiation of bevacizumab (day 15) and 1 month after initiation of bevacizumab (day 45). Arterialized venous blood samples will be collected during the imaging in order to measure radioactivity, blood metabolites, and the relationship between radiotracer uptake and tumor features such as blood-brain barrier (BBB) breakdown and tumor blood flow.
  In addition, we will explore the link between flow, permeability, and tumor temozolomide retention. These studies will be performed using our human simultaneous MRI-PET imaging camera.
  MRI-PET: - [11C] temozolomide for PET scan and
Arm/Group | TMZ-PET Scans/ MRI-PET Scan
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 62 [28 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 4
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Decrease in Median Tumor SUV
Description: Number of patients with a decrease in median tumor standard uptake value (SUV). Median tumor SUV was used as a marker of temozolomide uptake.
Time Frame: Day 15
Population: Tumor SUV measurements were only available for 8 patients
Measure: Count of Participants; unit: Participants
Arm/Group | TMZ-PET Scans/ MRI-PET Scan
Number analyzed (Participants) | 8
Participants | 6

ADVERSE EVENTS:
Time Frame: Up to day 42
Arm/Group | TMZ-PET Scans/ MRI-PET Scan
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 2/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TMZ-PET Scans/ MRI-PET Scan (N=12)
Wound Dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/30/NCT01987830/Prot_SAP_000.pdf